CLINICAL TRIAL: NCT00932334
Title: Culturally Sensitive Behavioral Interventions to Enhance Living Kidney Donation / Living Kidney Transplantation
Acronym: TALK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NA_00006752; R39OT07537
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Chronic Kidney Disease
Keywords: kidney; transplant; donation
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TALK Plus (Experimental): Participants receive and educational video and booklet about living kidney donation and meet with a social worker
  Interventions: Behavioral: TALK PLUS
- TALK Standard (Experimental): Participants receive and educational video and booklet about living kidney donation
  Interventions: Behavioral: TALK Standard
- Usual Care (Other): Participants receive their usual medical care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: TALK PLUS — Participants receive and educational video and booklet about living kidney donation and meet with a social worker
  Arms: TALK Plus
Behavioral: TALK Standard — Participants receive and educational video and booklet about living kidney donation
  Arms: TALK Standard
Behavioral: Usual Care — Participants receive their usual care
  Arms: Usual Care

SUMMARY:
Title: Culturally tailored behavioral interventions to enhance living kidney donation/living kidney transplantation Applicants: Johns Hopkins Medical Institutions, National Kidney Foundation of Maryland Principal Investigator: Neil R. Powe, MD, MPH, MBA Address: 2024 E. Monument Street, Suite 2-600, Baltimore, MD, 21205 Phone: 410-955-6953; Email: npowe@jhmi.edu; Fax: 410-955-0476 Rates of kidney donation have been largely stagnant for the past 10 years, resulting in large imbalances in numbers of persons on transplant waiting lists and the number of persons receiving kidney transplants. Slow improvement in donation and transplantation rates are exacerbated by ethnic/racial disparities in kidney transplants, in which minorities, particularly African Americans, are far less likely to receive deceased kidney transplants. Although living related kidney donation (LD) offers patients an opportunity to bypass many barriers contributing to disparities in kidney transplantation (e.g. waiting lists and immunological incompatibility issues), African Americans remain less likely to receive living related kidney transplants (LRT), further exacerbating disparities in transplant rates. Recent research demonstrates many ethnic minorities desire kidney transplantation, but rates of patient-physician and patient-family discussions regarding LD/LRT are suboptimal. Compared to Whites, African Americans have also been shown to have disproportionately greater rates of culture-specific concerns (such as mistrust in health care) that could impede them from seeking important medical therapies. It is unknown whether culturally tailored behavioral interventions to enhance patient/family decision-making regarding LD/LRT before the onset of end stage renal disease could improve rates of LD/LRT or could narrow racial disparities in the receipt of transplantation. The primary goal of this proposal is a) to use focus group methodology to develop culturally tailored educational materials for patients/families considering LD/LRT and b) to perform a randomized controlled trial to test the effectiveness of a culturally tailored social-worker led intervention (using established behavioral problem-solving therapeutic techniques) in enhancing rates of family communication, donor evaluations, and transplantation. The substantial experience of our consortium, including the National Kidney Foundation of Maryland and the Johns Hopkins Medical Institutions (Welch Center and the Medical Surgical Transplant Services in the School of Medicine), in the evaluation/ implementation of donor/recipient educational programs as well as the conduct of behavioral, epidemiologic and interventional studies related to donor/recipient health and psychology provides a strong foundation for the conduct of this study.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 70 with stage IV or stage V (non-dialysis dependent) chronic kidney disease

Exclusion Criteria:

* No evidence of cancer within 2 years prior to recruitment date
* No evidence of stage IV congestive heart failure
* No evidence of end-stage liver disease
* No evidence of unstable coronary artery disease
* No evidence of pulmonary hypertension
* No evidence of severe peripheral vascular disease
* No history of HIV
* No chronic (debilitating) infections
* No prior kidney transplant
* No prior completion of transplant evaluation process
* No prior dialysis treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
enhancing rates of family communication, donor evaluations, and transplantation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Leigh E Boulware, MD,MPH, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416
- [Derived] Boulware LE, Hill-Briggs F, Kraus ES, Melancon JK, Falcone B, Ephraim PL, Jaar BG, Gimenez L, Choi M, Senga M, Kolotos M, Lewis-Boyer L, Cook C, Light L, DePasquale N, Noletto T, Powe NR. Effectiveness of educational and social worker interventions to activate patients' discussion and pursuit of preemptive living donor kidney transplantation: a randomized controlled trial. Am J Kidney Dis. 2013 Mar;61(3):476-86. doi: 10.1053/j.ajkd.2012.08.039. Epub 2012 Oct 22. PMID 23089512
- [Derived] Boulware LE, Hill-Briggs F, Kraus ES, Melancon JK, McGuire R, Bonhage B, Senga M, Ephraim P, Evans KE, Falcone B, Troll MU, Depasquale N, Powe NR. Protocol of a randomized controlled trial of culturally sensitive interventions to improve African Americans' and non-African Americans' early, shared, and informed consideration of live kidney transplantation: the Talking About Live Kidney Donation (TALK) Study. BMC Nephrol. 2011 Jul 8;12:34. doi: 10.1186/1471-2369-12-34. PMID 21736762